CLINICAL TRIAL: NCT02871882
Title: Effect of Delayed-Release Bile Acid on Insulin Sensitivity, Gastric Emptying and Body Weight in Overweight or Obese Patients With Type 2 Diabetes Mellitus
Brief Title: Ox Bile- Conjugated Bile Acids Sodium in Type II Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Satiogen Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Andres J. Acosta, M.D., Ph.D., PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-007765
Record Dates: First submitted 2016-08-10; First posted 2016-08-18 (Estimated); Results first posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Type 2 Diabetes Mellitus; Obese; Overweight
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ox bile extract (Active Comparator): Ox bile extract 500 mg tablets taken orally twice daily for 28 (+/- 4) days Gastric Emptying test, Waist and hip measurements, Mixed oral glucose tolerance test, Blood tests
  Interventions: Radiation: Gastric Emptying test; Other: Mixed Oral Glucose Tolerance test; Drug: Conjugated bile acids sodium
- Placebo (Placebo Comparator): Matching placebo tablets taken orally twice daily for 28 (+/- 4) days Gastric Emptying test, Waist and hip measurements, Mixed oral glucose tolerance test, Blood tests
  Interventions: Radiation: Gastric Emptying test; Other: Mixed Oral Glucose Tolerance test; Other: Placebo

INTERVENTIONS:
Radiation: Gastric Emptying test — participants eat a standardized meal labeled with radioactive markers (99mTc DTPA [diethylenetriaminepentaacetic acid] and In111 Chloride). They have scans taken at specific times after the meal to document the rate of gastric emptying.
Other: Mixed Oral Glucose Tolerance test — Participants eat a meal containing 63g glucose in 240mL (milliliters) of skim milk, 2 scrambled eggs, 50g Canadian bacon and one slice of bread. Blood samples are taken prior to and for 6 hours after the meal at specific time points.
Drug: Conjugated bile acids sodium — 500 mg tablets taken orally twice daily for 28 (+/- 4) days
  Other Names: Ox Bile extract
  Arms: Ox bile extract
Other: Placebo — Placebo tablets taken orally twice daily for 28 (+/- 4) days
  Arms: Placebo

SUMMARY:
To study the effect of an ileocolonic formulation of ox bile extract on insulin sensitivity, postprandial glycemia and incretin levels, gastric emptying, body weight and fasting serum FGF-19 (fibroblast growth factor) levels in overweight or obese type 2 diabetic subjects on therapy with DPP4 (dipeptidyl peptidase-4) inhibitors (e.g. sitagliptin) alone or in combination with metformin.

DETAILED DESCRIPTION:
This is a single-center, placebo-controlled, parallel-group, single dose, randomized, controlled trial. Participants will receive 28 days (+/- 4 days) of treatment to study the effect of delayed (ileocolonic)-release ox bile extract 500 mg BID (twice daily) on insulin sensitivity, gastric emptying of liquids and solids (measured by scintigraphy) and weight loss I overweight and obese type 2 diabetic subjects. Participants will be receiving therapy with DPP4 inhibitors alone or in combination with metformin. Blood samples will be collected at defined times to measure glycemia, FGF-19 and incretins (GLP-1 [glucagon-like peptide-1], OXM [oxyntomodulin], PYY 3-36 [peptide YY]) fasting levels and responses to the meal.

ELIGIBILITY:
Inclusion criteria:

1. Overweight or obese subjects with BMI > 30 kg/m2 with type 2 diabetes mellitus taking DPP4 inhibitors alone or in combination with metformin.
2. Women of childbearing potential will have a negative pregnancy test before initiation of medication and within 48 hours of receiving radioisotope.

Exclusion criteria:

1. Structural of metabolic diseases/conditions that affect the gastrointestinal system, or functional gastrointestinal disorders.
2. Irritable bowel syndrome
3. Bristol stool type classification 4-7 per Bowel Disease questionnaire.
4. Subjects with other treatment for type 2 diabetes mellitus.
5. Subjects with HbA1c > 8%
6. Females who are pregnant or breastfeeding
7. Concomitant use of appetite suppressants, orlistat, phentermine-topiramate ER or lorcaserin.
8. Subjects who are not currently on treatment for cardiac, pulmonary, gastrointestinal, hepatic, renal, hematological, neurological, endocrine (other than type 2 diabetes mellitus), and unstable psychiatric disease.
9. Subjects who have donated blood or plasma in the past 8 weeks.
10. Subjects who have participated in another study within the past 30 days.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2017-10-18 (Actual); Study Completion 2017-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andres Acosta, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Calderon G, McRae A, Rievaj J, Davis J, Zandvakili I, Linker-Nord S, Burton D, Roberts G, Reimann F, Gedulin B, Vella A, LaRusso NF, Camilleri M, Gribble FM, Acosta A. Ileo-colonic delivery of conjugated bile acids improves glucose homeostasis via colonic GLP-1-producing enteroendocrine cells in human obesity and diabetes. EBioMedicine. 2020 May;55:102759. doi: 10.1016/j.ebiom.2020.102759. Epub 2020 Apr 25. PMID 32344198
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Ox Bile Extract: Ox bile extract 500 mg tablets taken orally twice daily for 28 (+/- 4) days Gastric Emptying test, Waist and hip measurements, Mixed oral glucose tolerance test, Blood tests
  Gastric Emptying test: participants eat a standardized meal labeled with radioactive markers (99mTc DTPA [diethylenetriaminepentaacetic acid] and In111 Chloride). They have scans taken at specific times after the meal to document the rate of gastric emptying.
  Mixed Oral Glucose Tolerance test: Participants eat a meal containing 63g glucose in 240mL (milliliters) of skim milk, 2 scrambled eggs, 50g Canadian bacon and one slice of bread. Blood samples are taken prior to and for 6 hours after the meal at specific time points.
  Conjugated bile acids sodium: 500 mg tablets taken orally twice daily for 28 (+/- 4) days
  Placebo: Placebo tablets taken orally twice daily for 28 (+/- 4) days
- Placebo: Matching placebo tablets taken orally twice daily for 28 (+/- 4) days Gastric Emptying test, Waist and hip measurements, Mixed oral glucose tolerance test, Blood tests
  Gastric Emptying test: participants eat a standardized meal labeled with radioactive markers (99mTc DTPA [diethylenetriaminepentaacetic acid] and In111 Chloride). They have scans taken at specific times after the meal to document the rate of gastric emptying.
  Mixed Oral Glucose Tolerance test: Participants eat a meal containing 63g glucose in 240mL (milliliters) of skim milk, 2 scrambled eggs, 50g Canadian bacon and one slice of bread. Blood samples are taken prior to and for 6 hours after the meal at specific time points.
  Conjugated bile acids sodium: 500 mg tablets taken orally twice daily for 28 (+/- 4) days
  Placebo: Placebo tablets taken orally twice daily for 28 (+/- 4) days
Period: Overall Study
Arm/Group | Ox Bile Extract | Placebo
Started | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ox Bile Extract | Placebo | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 60 [55 to 66] | 53 [45 to 65] | 57 [50 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 4 | 6 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 12 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change in Postprandial Glucose
Description: Measurement of the glucose concentration in the bloodstream 6 hours after eating a meal
Time Frame: baseline to 1 month
Measure: Mean (Inter-Quartile Range); unit: mmol/6hr
Arm/Group | Ox Bile Extract | Placebo
Number analyzed (Participants) | 11 | 12
mmol/6hr | -2803 [-5724 to 1098] | 629 [-4779 to 3814]
Statistical Analysis 1: Comparison: Ox Bile Extract vs Placebo; Test type: Superiority; p < 0.05, ANCOVA

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Ox Bile Extract | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 0/11 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-23): https://cdn.clinicaltrials.gov/large-docs/82/NCT02871882/Prot_SAP_000.pdf